CLINICAL TRIAL: NCT05470998
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of L-Arginine in Children Having Sickle Cell Disease With Increased Tricuspid Regurgitant Jet Velocity
Brief Title: L-Arginine in Children Having Sickle Cell Disease With Increased Tricuspid Regurgitant Jet Velocity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dalia Abdelhamid Gomaa, demonstrator at clinical pharmacy department, faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-Arginine 2021
Record Dates: First submitted 2022-07-17; First posted 2022-07-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Arginine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): this group will include 25 patients who will receive their standard therapy for 3 months
- L-Arginine group (Active Comparator): this group will include 25 patients who will receive L-Arginine 0.1-0.2 g/kg/day and their standard therapy for 3 months
  Interventions: Drug: L-Arginine

INTERVENTIONS:
Drug: L-Arginine — L-Arginine 1000 mg free form, rapid release capsules
  Arms: L-Arginine group

SUMMARY:
This study aims to investigate the possible efficacy and safety of L-Arginine in children having Sickle Cell Disease with increased Tricuspid Regurgitant Jet Velocity

ELIGIBILITY:
Inclusion Criteria:

* children having Sickle Cell Disease with increased Tricuspid Regurgitant Jet Velocity
* age 5-18 years

Exclusion Criteria:

* Another chronic hemolytic anemia.
* Patients with documented causes of pulmonary hypertension other than SCD.
* Allergy to L-arginine.
* Patients with Asthma.
* Hepatic dysfunction: serum Alanine Aminotransferase (ALT) > 3X upper value.
* Renal dysfunction: Creatinine level greater than or equal to 1.2 mg/dl.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
change in tricuspid regurgitant jet velocity (TRJV) detected by Color Doppler Echocardiography | 3 months
  patients will undergo Color Doppler Echocardiography to assess tricuspid regurgitant jet velocity (TRJV) at baseline and after 3 months

SECONDARY OUTCOMES:
change in serum level of N-terminal pro b-type natriuretic peptide (NT-pro-BNP) | 3 months
  Blood samples will be collected at baseline and after 3 months
change in serum level of L-Arginine | 3 months
  Blood samples will be collected at baseline and after 3 months
change in serum level of Asymmetric Dimethyl Arginine (ADMA) | 3 months
  Blood samples will be collected at baseline and after 3 months
change in serum level of Nitric Oxide | 3 months
  Blood samples will be collected at baseline and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: dalia A gomaa, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Other (Non U.s.), Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomaa DA, El-Haggar SM, El-Shanshory MR, El-Razaky O, El-Afify DR. Clinical Study to Evaluate the Possible Efficacy and Safety of L-Arginine in Children with Sickle Cell Disease and Increased Tricuspid Regurgitant Jet Velocity: a Randomized Controlled Trial. Paediatr Drugs. 2025 Sep;27(5):605-618. doi: 10.1007/s40272-025-00701-w. Epub 2025 Jun 17. PMID 40526198